CLINICAL TRIAL: NCT02822534
Title: the Pharmacokinetics,Pharmacodynamics,Safety and Tolerability Study Following Single and Multiple Dose of SP2086 in Type 2 Diabetes Patients
Brief Title: The Pharmacokinetics and Pharmacodynamics Study of Single and Multiple Dose of SP2086 in Type 2 Diabetes Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SP2086-113
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SP2086 50mg (Experimental): there were 3 groups in the study: 50mg ,100mg and 200mg ,each group including 8 Type 2 diabetes patients.All subjects were administrated the medicine at Day 1 and Day 5 to Day 9.During the test,collecting the blood samples were needed before and after taking medicine.
  Interventions: Drug: SP2086
- SP2086 100mg (Experimental): there were 3 groups in the study: 50mg ,100mg and 200mg ,each group including 8 Type 2 diabetes patients.All subjects were administrated the medicine at Day 1 and Day 5 to Day 9.During the test,collecting the blood samples were needed before and after taking medicine.
  Interventions: Drug: SP2086
- SP2086 200mg (Experimental): there were 3 groups in the study: 50mg ,100mg and 200mg ,each group including 8 Type 2 diabetes patients.All subjects were administrated the medicine at Day 1 and Day 5 to Day 9.During the test,collecting the blood samples were needed before and after taking medicine.
  Interventions: Drug: SP2086

INTERVENTIONS:
Drug: SP2086 — the study has 3 doses groups and the 24 subjects were administrated SP2086 50mg,100mg,200mg respectively.

SUMMARY:
SP2086 is a novel inhibitor of Dipeptide base peptidase 4, allows an insulin-independent approach to improve type 2 diabetes hyperglycemia. In this single-dose and multiple-dose study the investigators evaluated the safety, tolerability and PK/PD profiles of SP2086 in Type 2 Diabetes Patients .

ELIGIBILITY:
Inclusion Criteria:

* The patient has a definitive diagnosis of Type 2 Diabetes.
* BMI(a measure of a person's weight in relation to height)is between 19 and 30 kg/m2,and the weight is equal or greater than 50kg.
* Never use the antidiabetic or only use one type oral antidiabetic(except the insulin secretagogues agent).
* The patient never use insulin in 3 months of screening.
* Be willing to accept physical contraception.
* Sign the informed consents voluntarily and ensure to completed the study.

Exclusion Criteria:

* The value of fasting blood-glucose(FBG)>13.9mmol/L,or HbA1c>10.0%;
* Known allergy to SP2086 or any of the excipients of the formulation of SP2086;
* Type 1 diabetes,or Gestational diabetes,or other type diabetes;
* ever occured acute complications of diabetes such as diabetic ketoacidosis,high permeability syndrome or lactic acidosis.
* ever occured the severe hypoglycemia.
* History of chronic complication of diabetes(kidney disease,or retinopathy,neuropathy,or lower limb vascular lesion).
* The value of serum creatinine over the upper limit of normal range.
* ever occured myocardial infarction,acute coronary syndrome, transient ischemic attack.
* QTc interval>450ms(male) or >470ms(female) or have the history of cardiac insufficiency which the NYHA(New York Heart Association) class over I degree.
* have the history of hypertension,and not well control:SBP(Systolic Blood Pressure)>140 mmHg or DBP(Diastolic Blood Pressure)>90 mmHg.
* have the history of cancer.
* the value of ALT and/or AST was greater two times of upper limit of normal range,or the STB over the 1.5 times of upper limit of normal range.
* the B hepatitis surface antigen or hepatitis C antibody or syphilis antibody or HIV antibody was positive.
* had participated three or more clinical trial in one year or had participated one time clinical medicine in one month of screening.
* have the history of blood donation in 3 months of screening or received the blood transfusion in 1 months of screening.
* have the history of tobacco,alcohol or drug abuse.
* History of or current clinically significant medical illness as determined by the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SP2086 | up to Day 13
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of SP2086
The steady-state plasma concentration (Css) of SP2086 | up to Day 13
  Css (a measure of the body's exposure to SP2086) will be compared before and after administration of multiple doses of SP2086
The maximum plasma concentration (Cmax) of SP2086 acid | up to Day 13
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of SP2086
The steady-state plasma concentration (Css) of SP2086 acid | up to Day 13
  Css (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086
The maximum urine concentration (Cmax) of SP2086 | up to Day 13
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of SP2086
The steady-state urine concentration (Css) of SP2086 | up to Day 13
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of SP2086
The maximum urine concentration (Cmax) of SP2086 acid | up to Day 13
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of SP2086
The steady-state urine concentration (Css) of SP2086 acid | up to Day 13
  Css (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 13

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hosital of Jilin University, Changchun, Jilin, China